CLINICAL TRIAL: NCT06218927
Title: The Effect of Autologous Hematopoietic Stem Cell Transplantation on the Lower Urinary Tract Function Related Quality of Life in Multiple Sclerosis Patients
Brief Title: The Effect of Autologous Hematopoietic Stem Cell Transplantation on the Lower Urinary Tract Function Related to QoL in MS Patients
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-URO-RS-2023
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis; Lower Urinary Tract Symptoms
Keywords: Multiple Sclerosis; Lower Urinary Tract Symptoms; Autologous Hematopoietic Stem Cell Transplantation; Disease-Modifying Therapy; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autologous hematopoietic stem cell transplantation (AHSCT): Patients who underwent autologous hematopoietic stem cell transplantation (AHSCT).
  Interventions: Other: QoL monitoring
- Disease-modifying therapy: Patients who undergo disease-modifying therapy - standard treatment.
  Interventions: Other: QoL monitoring

INTERVENTIONS:
Other: QoL monitoring — QoL questionnaire

SUMMARY:
Academic research project monitoring the effect of Autologous Hematopoietic Stem Cell Transplantation (AHSCT) on multiple sclerosis-associated lower urinary tract symptoms.

DETAILED DESCRIPTION:
An observational study (academic research project) monitoring the effect of autologous hematopoietic stem cell transplantation (AHSCT) in patients with multiple sclerosis (MS) on lower urinary tract symptoms occurrence. The main goal is to observe the influence of this treatment modality on changes in the quality of life. Secondary endpoints are the changes in the urodynamic parameters and lower urinary tract occurrence. The investigators assume the inclusion of a minimum of 20 patients with AHSCT and 20 patients in the control group with other disease-modifying therapy (DMT).

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male and female) aged 18 and over
* Subjects with signed informed consent
* Subjects able to undergo examination according to the protocol
* Patients indicated by neurologists to perform AHSCT or treated with the closest similar disease-modifying therapy (control group)

Exclusion Criteria:

* Subjects with a history of bladder cancer
* Subjects after previous pelvic radiotherapy
* Subjects with evidence of microscopic or macroscopic hematuria
* Subjects with a history of bladder reconstruction (augmentation cystoplasty, catheterizable stoma), subjects after cystectomy
* Treatment with botulinum toxin injection into the bladder wall in the last 12 months
* Patients in whom the pharmacological treatment of the lower urinary tract has not been stable in the last 3 months and is being adjusted
* Patients whose lower urinary tract symptoms are not stable for at least 3 months
* Patients with a permanent catheter
* Patients with recurrent symptomatic lower urinary tract infections - 3 or more episodes of infection in the last 12 months
* Subjects with tubal urine screening-proven bacteriuria
* Patients with acute lower urinary tract inflammation at baseline
* Subjects with painful bladder syndrome
* Patients after sacral neuromodulation
* Patients with severe pelvic organ prolapse
* Patients after radical pelvic surgery
* Patients with a life expectancy of less than 5 years at the time of inclusion in the study
* Lactating women, pregnant women, women trying to get pregnant, or sexually active women without a tendency to use safe contraception (hormonal-based oral contraceptives, injectable contraception, hormonally active implants, sexual abstinence, vasectomy in a partner)
* Subjects who participated in another study in the previous 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis referred for HSCT or referred for other DMT.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
QoL changes associated with MS treatment | 30 months
  The overall score from the baseline to the end of follow-up will be calculated, using the Qualiveen questionnaire. The 30-item Qualiveen is a specific health-related quality-of-life questionnaire for urinary disorders in patients with neurological conditions.

SECONDARY OUTCOMES:
Neurogenic Bladder Symptom Score (NBSS) | 30 months
  The change in lower urinary tract symptoms will be measured by the NBSS score, from baseline to the end of follow-up. The Neurogenic Bladder Symptom Score (NBSS) (24-item) is a freely available, self-administered, questionnaire that assesses urinary symptoms and bladder-related consequences in patients with acquired or congenital neurogenic bladder dysfunction as a result of spinal cord injury, multiple sclerosis, and spinal bifida.
Patient satisfaction (PGI-I) | 30 months
  Patient satisfaction associated with the treatment of multiple sclerosis will be monitored using the PGI-I tool (Patient Global Impression of Improvement) from baseline to the end of follow-up. The PGI-I is a global index that may be used to rate the response of a condition to a therapy (transition scale).

CONTACTS AND LOCATIONS:
Overall Officials: Radek Paus Sýkora, MD, Principal Investigator — University Hospital Ostrava; Jan Krhut, prof.,MD,PhD, Study Director — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Cohen RA, Kessler HR, Fischer M. The Extended Disability Status Scale (EDSS) as a predictor of impairments of functional activities of daily living in multiple sclerosis. J Neurol Sci. 1993 Apr;115(2):132-5. doi: 10.1016/0022-510x(93)90215-k. PMID 8482974
- [Background] Lublin FD, Reingold SC. Defining the clinical course of multiple sclerosis: results of an international survey. National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. Neurology. 1996 Apr;46(4):907-11. doi: 10.1212/wnl.46.4.907. PMID 8780061
- [Background] Doshi A, Chataway J. Multiple sclerosis, a treatable disease. Clin Med (Lond). 2016 Dec;16(Suppl 6):s53-s59. doi: 10.7861/clinmedicine.16-6-s53. PMID 27956442
- [Background] Henze T, Rieckmann P, Toyka KV; Multiple Sclerosis Therapy Consensus Group of the German Multiple Sclerosis Society. Symptomatic treatment of multiple sclerosis. Multiple Sclerosis Therapy Consensus Group (MSTCG) of the German Multiple Sclerosis Society. Eur Neurol. 2006;56(2):78-105. doi: 10.1159/000095699. Epub 2006 Sep 8. PMID 16966832
- [Background] de Seze M, Ruffion A, Denys P, Joseph PA, Perrouin-Verbe B; GENULF. The neurogenic bladder in multiple sclerosis: review of the literature and proposal of management guidelines. Mult Scler. 2007 Aug;13(7):915-28. doi: 10.1177/1352458506075651. Epub 2007 Mar 15. PMID 17881401
- [Background] Schneider MP, Tornic J, Sykora R, Abo Youssef N, Mordasini L, Krhut J, Chartier-Kastler E, Davies M, Gajewski J, Schurch B, Bachmann LM, Kessler TM. Alpha-blockers for treating neurogenic lower urinary tract dysfunction in patients with multiple sclerosis: A systematic review and meta-analysis. A report from the Neuro-Urology Promotion Committee of the International Continence Society (ICS). Neurourol Urodyn. 2019 Aug;38(6):1482-1491. doi: 10.1002/nau.24039. Epub 2019 May 16. PMID 31099113
- [Background] Panicker JN. Neurogenic Bladder: Epidemiology, Diagnosis, and Management. Semin Neurol. 2020 Oct;40(5):569-579. doi: 10.1055/s-0040-1713876. Epub 2020 Oct 16. PMID 33065745
- [Background] Alsaid B, Moszkowicz D, Peschaud F, Bessede T, Zaitouna M, Karam I, Droupy S, Benoit G. Autonomic-somatic communications in the human pelvis: computer-assisted anatomic dissection in male and female fetuses. J Anat. 2011 Nov;219(5):565-73. doi: 10.1111/j.1469-7580.2011.01416.x. Epub 2011 Jul 22. PMID 21781094
- [Background] Abello A, Das AK. Electrical neuromodulation in the management of lower urinary tract dysfunction: evidence, experience and future prospects. Ther Adv Urol. 2018 Feb 22;10(5):165-173. doi: 10.1177/1756287218756082. eCollection 2018 May. PMID 29623108
- [Background] Michel MC, Sand C. Effect of pre-contraction on beta-adrenoceptor-mediated relaxation of rat urinary bladder. World J Urol. 2009 Dec;27(6):711-5. doi: 10.1007/s00345-009-0416-y. PMID 19449014
- [Background] Cartwright R, Panayi D, Cardozo L, Khullar V. Reliability and normal ranges for the Patient's Perception of Intensity of Urgency Scale in asymptomatic women. BJU Int. 2010 Mar;105(6):832-6. doi: 10.1111/j.1464-410X.2009.08846.x. Epub 2009 Oct 10. PMID 19818081
- [Background] Schafer W, Abrams P, Liao L, Mattiasson A, Pesce F, Spangberg A, Sterling AM, Zinner NR, van Kerrebroeck P; International Continence Society. Good urodynamic practices: uroflowmetry, filling cystometry, and pressure-flow studies. Neurourol Urodyn. 2002;21(3):261-74. doi: 10.1002/nau.10066. PMID 11948720
- [Background] Dicuio M, Pomara G, Menchini Fabris F, Ales V, Dahlstrand C, Morelli G. Measurements of urinary bladder volume: comparison of five ultrasound calculation methods in volunteers. Arch Ital Urol Androl. 2005 Mar;77(1):60-2. PMID 15906795
- [Background] Bonniaud V, Bryant D, Parratte B, Guyatt G. Qualiveen, a urinary-disorder specific instrument: 0.5 corresponds to the minimal important difference. J Clin Epidemiol. 2008 May;61(5):505-10. doi: 10.1016/j.jclinepi.2007.06.008. Epub 2008 Jan 7. PMID 18394545
- [Background] Welk B, Morrow S, Madarasz W, Baverstock R, Macnab J, Sequeira K. The validity and reliability of the neurogenic bladder symptom score. J Urol. 2014 Aug;192(2):452-7. doi: 10.1016/j.juro.2014.01.027. Epub 2014 Feb 8. PMID 24518764